CLINICAL TRIAL: NCT07283237
Title: Enhancing Medial Knee Pain Rehabilitation : A Clinical Trial On The Effectiveness Of Blood Flow Restriction In Combination With Targeted Exercises For Adult With Varus Deformity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam ibrahim, Physical Therapy Research Fellow, Assiut University, EGYPT, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-2025-300646
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis (Mild to Moderate, Medial Compartment)
Keywords: Medial knee pain; Varus knee deformity; Blood flow restriction (BFR)
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - Targeted Exercise Program (Active Comparator): Participants in the control group will perform a specific targeted exercise program focusing on hip adductors, abductors, internal rotators, and knee extensors. Exercises will be performed at moderate intensity without any blood flow restriction. The program aims to improve lower limb alignment, muscle balance, and functional performance through conventional strengthening exercises.
  Interventions: Behavioral: Targeted Exercise Program
- Intervention Group - Blood Flow Restriction (BFR) with Targeted Exercise Program (Experimental): Participants in the intervention group will perform the same targeted exercise program (hip adductors, abductors, internal rotators, and knee extensors) combined with Blood Flow Restriction (BFR) using a Smart Tools Plus (LLC, USA) pneumatic cuff applied to the proximal thigh.
  Cuff pressure will be set individually at 40-80% of limb occlusion pressure (LOP), maintained during exercise sets and released during 1-minute rest intervals. The intervention aims to enhance muscle strength and function while minimizing joint stress and pain.
  Interventions: Device: Blood Flow Restriction (BFR) Training with Targeted Exercise Program

INTERVENTIONS:
Behavioral: Targeted Exercise Program — A structured therapeutic exercise program designed to strengthen the hip adductors, abductors, internal rotators, and knee extensors. The program focuses on improving muscular balance, lower limb alignment, and functional performance in active adults with medial knee pain and varus deformity. Exercises are performed under therapist supervision at moderate intensity without blood flow restriction. This program serves as the control intervention.
  Arms: Control Group - Targeted Exercise Program
Device: Blood Flow Restriction (BFR) Training with Targeted Exercise Program — Participants perform the same targeted exercise program combined with Blood Flow Restriction (BFR) training using a Smart Tools Plus (LLC, USA) pneumatic cuff system applied to the proximal thigh.
  Cuff pressure is individually set at 40-80% of the limb occlusion pressure (LOP), maintained during exercise sets and released during rest intervals (1 minute between sets). The intervention aims to enhance muscle strength and hypertrophy while reducing joint load and pain, providing an effective rehabilitation approach for adults with medial knee pain and varus deformity.
  Arms: Intervention Group - Blood Flow Restriction (BFR) with Targeted Exercise Program

SUMMARY:
Medial knee pain is common in active adults with varus knee alignment and can limit daily and sports activities. Standard physiotherapy can reduce pain and improve function, but strength gains may be suboptimal when patients cannot tolerate high loading due to pain. Blood flow restriction (BFR) training allows muscle strength and hypertrophy improvements at low external loads by partially restricting limb blood flow, thereby reducing joint stress. Although BFR has shown benefits in people with knee osteoarthritis, its effectiveness for medial knee pain associated with varus deformity is not well established.

This randomized controlled trial will investigate whether adding BFR to a targeted strengthening program provides superior outcomes compared with the same exercise program alone in active adults with medial knee pain and mild to moderate varus alignment. Approximately 80 participants aged 30-55 years with BMI 18-25, medial knee pain, Kellgren-Lawrence grade 1-3 osteoarthritis, and Hip-Knee-Ankle angle between >2° and ≤10° varus will be recruited from an outpatient setting. Participants will be randomly assigned (1:1) to either a specific exercise program (hip adductors/abductors, internal rotators, and knee extensors) or the same program performed with BFR using a pneumatic thigh cuff set at 40-80% limb occlusion pressure. Outcomes, including the Oxford Knee Score (primary), lower-extremity function, pain, quality of life, muscle strength, radiographic alignment, and relapse rates over 12 months, will be assessed at baseline and multiple follow-up points by blinded assessors.

DETAILED DESCRIPTION:
Medial knee pain in the presence of varus malalignment is a frequent clinical presentation in active adults and is strongly associated with increased medial compartment loading, progressive cartilage degeneration, and an elevated risk of symptomatic knee osteoarthritis. In patients with persistent symptoms and structural progression, realignment surgery such as high tibial osteotomy (HTO) is considered when the hip-knee-ankle (HKA) angle exceeds approximately 3° of varus and is often recommended at 5°-6° or more of symptomatic varus in relatively young, active individuals with preserved lateral compartment cartilage. In this context, mild, moderate, and severe varus deformities have been described in the literature as roughly 3°-5°, 6°-8°, and ≥9° of varus alignment, respectively. For many patients, however, there is a substantial window in which optimized conservative management could delay or possibly reduce the need for surgical realignment while improving pain and function.

Conventional physiotherapy and strengthening programs for medial knee pain and early knee osteoarthritis typically emphasize quadriceps and general lower-limb strengthening, flexibility, and neuromuscular training. These approaches can reduce pain and improve function but may not always achieve optimal muscle adaptation because patients often cannot tolerate high-load resistance exercise due to joint pain or fear of aggravating symptoms. As a result, clinicians are frequently constrained to suboptimal loading intensities, which may limit gains in strength and neuromuscular control that are needed to better support the varus knee and potentially reduce medial compartment load during everyday and sports activities.

Blood flow restriction (BFR) training has emerged as a promising adjunct in musculoskeletal rehabilitation, enabling meaningful improvements in muscle strength and hypertrophy at relatively low external loads. By applying a pneumatic cuff to partially restrict venous outflow while maintaining arterial inflow, BFR produces a metabolic and mechanical environment that mimics high-load training, but with considerably less joint stress. This is particularly relevant in populations with painful knee osteoarthritis or varus deformity, where high-load training is often poorly tolerated. Recent trials in knee osteoarthritis populations suggest that low-load BFR-enhanced exercise can lead to clinically important improvements in pain, muscle strength, and quality of life compared with similar exercise performed without BFR. However, the specific role of BFR in active adults with medial knee pain and varus malalignment has not been adequately explored.

This randomized controlled trial is designed to compare a targeted lower-limb strengthening and neuromuscular program alone with the same program combined with BFR in active adults with medial knee pain, mild to moderate varus deformity, and radiographic knee osteoarthritis (Kellgren-Lawrence grade 1-3). Eligible participants will be recruited from an outpatient physical therapy setting and will meet predefined clinical and radiographic criteria (detailed in the Eligibility section), including age range, body mass index, degree of varus malalignment on long-leg radiographs, and activity level. The sample size was determined a priori using G*Power to detect a moderate effect size in repeated-measures analyses with two groups and multiple time points, with additional allowance for attrition to yield an enrollment target of approximately 80 participants.

Participants will be allocated in a 1:1 ratio to either a control group receiving a specific exercise program or an experimental group performing the same exercises with the addition of BFR. The specific exercise program is designed to address key muscle groups that contribute to frontal-plane control and dynamic alignment of the lower limb, with a particular focus on the hip adductors, abductors, internal rotators, and knee extensors. Exercises will be delivered in a progressive manner over a 6-week supervised intervention period in the outpatient clinic, with standardized progression criteria and an accompanying home-exercise component to reinforce clinic-based training.

In the BFR group, a commercially available pneumatic cuff system (Smart Tools Plus, LLC, USA) will be placed on the proximal thigh of the affected limb during selected strengthening exercises. Cuff pressure will be individualized using limb occlusion pressure (LOP) testing, and exercise sessions will be conducted at a percentage of LOP (e.g., 40-80%), consistent with published safety and efficacy recommendations for low-load BFR training. The cuff will be inflated during each exercise set and deflated during rest intervals to minimize discomfort and reduce the risk of adverse events. Participants will be monitored throughout each session for signs of intolerance or complications, such as disproportionate pain, numbness, dizziness, or skin discoloration, and predefined criteria will guide modification or discontinuation of BFR as needed.

Outcome assessments will be performed at baseline and at multiple follow-up time points after the intervention, including early post-treatment and longer-term follow-ups. The primary endpoint of the trial is improvement in knee-specific pain and function as captured by a validated patient-reported outcome measure. Secondary endpoints include changes in general lower-extremity function, pain intensity, health-related quality of life, objective measures of hip muscle strength using a handheld dynamometer, and radiographic parameters of lower-limb mechanical alignment, as well as the incidence of symptom relapses over a 12-month observation period. All clinical and radiographic outcome measures will be obtained by assessors who are blinded to group allocation to reduce measurement bias.

Statistical analyses will compare trajectories of change between the two intervention arms over time, using repeated-measures approaches appropriate for continuous outcomes and suitable tests for categorical data. The primary analysis will follow the intention-to-treat principle, with additional per-protocol or sensitivity analyses as appropriate. By systematically evaluating the additive effect of BFR on top of a targeted strengthening program in this specific population, the trial aims to determine whether BFR-enhanced exercise yields superior outcomes in pain, function, muscle strength, and alignment compared with exercise alone, potentially informing more effective conservative treatment strategies for active adults with varus-related medial knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 55 years
* Body Mass Index (BMI) between 18 and 25
* Presence of medial knee pain
* Mild to moderate varus deformity confirmed via X-Ray Long Film (2° < HKA ≤ 10°) (4)(4)(5)
* Kellgren and Lawrence classification of osteoarthritis (grades 1-3) (6):
* Grade 1 (doubtful): doubtful joint space narrowing and possible osteophytic lipping
* Grade 2 (minimal): definite osteophytes and possible joint space narrowing
* Grade 3 (moderate): moderate multiple osteophytes, definite narrowing of joint space, some sclerosis and possible deformity of bone ends
* Active adults (based on REFA work classification)

Exclusion Criteria:

* BMI > 25
* History of knee surgery
* Any contraindication to exercise or BFR, including:
* History of deep vein thrombosis (DVT)
* Uncontrolled hypertension
* Peripheral vascular disease
* Pregnancy
* Other significant musculoskeletal or neurological conditions affecting lower extremity function (e.g., hip osteoarthritis, rheumatoid arthritis, peripheral neuropathy)

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) | Baseline, 6 weeks (post-intervention), 3 months, and 6 months follow-up.
  The Oxford Knee Score (OKS) is a validated 12-item questionnaire designed to assess knee function and pain during daily activities. Each item is scored from 0 to 4, with higher total scores indicating better knee function and reduced pain. It evaluates activities such as walking, climbing stairs, and rising from a chair, reflecting the participant's perceived level of recovery and functional ability.

SECONDARY OUTCOMES:
Lower Extremity Functional Scale (LEFS) | Baseline, 6 weeks, 3 months, and 6 months follow-up.
  The LEFS is a 20-item self-reported questionnaire used to assess functional status in individuals with lower limb musculoskeletal conditions. Each item is scored from 0 (extreme difficulty) to 4 (no difficulty), with higher scores indicating better functional performance.
Short Form-36 (SF-36) Quality of Life Questionnaire | Baseline, 6 weeks, 3 months, and 6 months follow-up.
  The SF-36 is a standardized tool for assessing health-related quality of life across eight domains including physical functioning, bodily pain, vitality, and general health perception. Scores are transformed into a 0-100 scale, with higher scores indicating better quality of life.
Numerical Pain Rating Scale (NPRS) | Baseline, 6 weeks, 3 months, and 6 months follow-up.
  The NPRS is a subjective measure of pain intensity rated by participants on a scale from 0 (no pain) to 10 (worst imaginable pain). It captures current, best, and worst pain levels to assess changes in pain perception following intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Indications and clinical outcomes of High Tibial Osteotomy: A literature review. Available from: https://meddocsonline.org/journal-of-orthopedics-and-muscular-system/indications-and-clinical-outcomes-of-high-tibial-osteotomy-a-literature-review.html?utm_source=chatgpt.com
- [Background] Feucht MJ, Winkler PW, Mehl J, Bode G, Forkel P, Imhoff AB, Lutz PM. Isolated high tibial osteotomy is appropriate in less than two-thirds of varus knees if excessive overcorrection of the medial proximal tibial angle should be avoided. Knee Surg Sports Traumatol Arthrosc. 2021 Oct;29(10):3299-3309. doi: 10.1007/s00167-020-06166-3. Epub 2020 Jul 20. PMID 32691093
- [Background] Pipino G, Indelli PF, Tigani D, Maffei G, Vaccarisi D. Opening-wedge high tibial osteotomy: a seven - to twelve-year study. Joints. 2016 Jun 13;4(1):6-11. doi: 10.11138/jts/2016.4.1.006. eCollection 2016 Jan-Mar. PMID 27386441
- [Background] Elbardesy H, McLeod A, Ghaith HS, Hakeem S, Housden P. Outcomes of double level osteotomy for osteoarthritic knees with severe varus deformity. A systematic review. SICOT J. 2022;8:7. doi: 10.1051/sicotj/2022009. Epub 2022 Apr 1. PMID 35363133
- [Background] Kohn MD, Sassoon AA, Fernando ND. Classifications in Brief: Kellgren-Lawrence Classification of Osteoarthritis. Clin Orthop Relat Res. 2016 Aug;474(8):1886-93. doi: 10.1007/s11999-016-4732-4. Epub 2016 Feb 12. No abstract available. PMID 26872913
- [Background] Bennell KL, Bowles KA, Wang Y, Cicuttini F, Davies-Tuck M, Hinman RS. Higher dynamic medial knee load predicts greater cartilage loss over 12 months in medial knee osteoarthritis. Ann Rheum Dis. 2011 Oct;70(10):1770-4. doi: 10.1136/ard.2010.147082. Epub 2011 Jul 7. PMID 21742637
- [Background] Zeng CY, Zhang ZR, Tang ZM, Hua FZ. Benefits and Mechanisms of Exercise Training for Knee Osteoarthritis. Front Physiol. 2021 Dec 16;12:794062. doi: 10.3389/fphys.2021.794062. eCollection 2021. PMID 34975542